CLINICAL TRIAL: NCT02638428
Title: Genomics-Based Target Therapy for Children With Relapsed or Refractory Malignancy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-08-008
Record Dates: First submitted 2015-11-29; First posted 2015-12-23 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Relapsed Pediatric Solid Tumor; Refractory Pediatric Solid Tumor; Relapsed Pediatric AML; Refractory Pediatric AML
MeSH Terms: interventions — Ifosfamide; Carboplatin; Etoposide; fludarabine; Cytarabine; pazopanib; Sorafenib; Axitinib; Crizotinib; Dasatinib; Erlotinib Hydrochloride; Everolimus; Imatinib Mesylate; ruxolitinib; vandetanib; Vemurafenib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Refractory/relapsed solid tumor or AML (Experimental): Conventional chemotherapy (Ifosfamide carboplatin etoposide for solid tumor and fludarabine cytarabine for AML) with matched single-targeted agent (axitinib, crizotinib, dasatinib, erlotinib, everolimus, imatinib, pazopanib, ruxolitinib, sorafenib, vandetanib, vemurafenib, or trastuzumab) or multi-targeted receptor tyrosine kinase inhibitor (pazopanib or sorafenib) according to the result of CancerSCAN™
  Interventions: Procedure: CancerSCAN™; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: Fludarabine; Drug: Cytarabine; Drug: Pazopanib; Drug: Sorafenib; Drug: Axitinib; Drug: Crizotinib; Drug: Dasatinib; Drug: Erlotinib; Drug: Everolimus; Drug: Imatinib; Drug: Ruxolitinib; Drug: Vandetanib; Drug: Vemurafenib; Drug: Trastuzumab

INTERVENTIONS:
Procedure: CancerSCAN™ — Targeted deep sequencing
Drug: Ifosfamide
Drug: Carboplatin
Drug: Etoposide
Drug: Fludarabine
Drug: Cytarabine
Drug: Pazopanib
Drug: Sorafenib
Drug: Axitinib
Drug: Crizotinib
Drug: Dasatinib
Drug: Erlotinib
Drug: Everolimus
Drug: Imatinib
Drug: Ruxolitinib
Drug: Vandetanib
Drug: Vemurafenib
Drug: Trastuzumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and feasibility of combination chemotherapy with target agents according to the result of targeted deep sequencing in pediatric patients with relapsed/refractory solid tumor or AML.

DETAILED DESCRIPTION:
Outcome of pediatric cancer has been improved substantially over the past few decades, but the prognosis of relapsed/refractory pediatric cancer still remains poor. Advances in genomic technologies have improved the ability to detect diverse somatic and germline genomic aberrations of cancer patients, and it has been incorporated in the clinical management of cancer.

Samsung Genomic Institute developed a targeted next-generation sequencing (NGS) platform, CancerSCAN™, which can detect clinically significant genomic aberrations of tumors. In this study, tumor samples of refractory/relapsed pediatric cancer patients will be tested with CancerSCAN™ and the patients will receive combination chemotherapy with matched single-targeted agent or multi-targeted receptor tyrosine kinase inhibitor according to the result of CancerSCAN™.

I. Relapsed/refractory solid tumor

* Perform CancerSCAN™ at enrollment
* Conventional chemotherapy (ifosfamide, carboplatin, etoposide) with matched single-targeted agent (axitinib, crizotinib, dasatinib, erlotinib, everolimus, imatinib, pazopanib, ruxolitinib, sorafenib, vandetanib, vemurafenib, or trastuzumab) or multi-targeted receptor tyrosine kinase inhibitor (pazopanib or sorafenib) according to the result of CancerSCAN™

II. Relapsed/refractory AML

* Perform CancerSCAN™ at enrollment
* Conventional chemotherapy (fludarabine, cytarabine) with matched single-targeted agent (axitinib, crizotinib, dasatinib, erlotinib, everolimus, imatinib, pazopanib, ruxolitinib, sorafenib, vandetanib, vemurafenib, or trastuzumab) or multi-targeted receptor tyrosine kinase inhibitor (pazopanib or sorafenib) according to the result of CancerSCAN™

ELIGIBILITY:
Inclusion Criteria:

* Under 18 years of age at initial diagnosis
* Patients with refractory/relapsed solid tumor or AML (Solid tumor: Stable or progressive disease after 1st-line treatment or relapse; AML: Persistence after 2 cycles of induction chemotherapy or relapse)
* Patient with tumor sample which is adequate for targeted deep sequencing

Exclusion Criteria:

* Patients who had salvage chemotherapy previously
* Patients with organ dysfunction as follows (creatinine elevation ≥ 3 x upper limit of normal (ULN), ejection fraction <40%, significant arrhythmia or conduction disturbance)
* Patients who are not eligible to have scheduled treatment due to the other significant impaired organ function
* Patients whose tumor samples are not sufficient for targeted deep sequencing
* Pregnant or nursing women

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-12; Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Rate of event free survival | Up to 5 years
  Event is defined as relapse, disease progression or treatment-related mortality.

SECONDARY OUTCOMES:
Rate of treatment-related adverse events as assessed by CTCAE v4.0 | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Sung, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea